CLINICAL TRIAL: NCT05335941
Title: A Phase 2 Study to Evaluate the Triplet Combination of Pemetrexed Plus AB928 (Etrumadenant) + AB122 (Zimberelimab) in Patients With Previously Treated Advanced or Metastatic MTAP Deficient Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0774; NCI-2022-02708 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-03-24; First posted 2022-04-20 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Urothelial Carcinoma; Metastatic Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasm Metastasis | interventions — Pemetrexed; zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pemetrexed Plus AB928 (Etrumadenant) Plus AB122 (Zimberelimab) (Experimental): All patients will receive combination therapy of pemetrexed and ZIMBERELIMAB (AB122) intravenously every 3 weeks as well as ETRUMADENANT (AB928) orally daily.
  Interventions: Drug: Pemetrexed; Drug: Zimberelimab; Drug: Etrumadenant

INTERVENTIONS:
Drug: Pemetrexed — Given by vein (IV)
  Other Names: LY23151; Alimta®; MTA; Multitargeted Antifolate; NSC-698037
Drug: Zimberelimab — Given by vein (IV)
  Other Names: AB122
Drug: Etrumadenant — Given by PO
  Other Names: AB928; Etruma

SUMMARY:
This is a Phase 2 open-label, single-arm trial for patients with MTAP-deficient advanced urothelial cancer who had received prior immunotherapy. This is a single site study at the University of Texas MD Anderson Cancer Center. This study will allow patients in second line of treatment for advanced urothelial ca or beyond. All patients must have been previously treated with immune checkpoint inhibitor (ICI) therapy as per current standard of care.

DETAILED DESCRIPTION:
Objectives:

Primary Objectives:

* To evaluate the safety and tolerability of the triplet combination regimen.
* To evaluate the clinical activity of the triplet combination regimen.

Secondary Objectives:

* To explore the biological changes in MTAP-deficient UC tumor microenvironment including peripheral T-cells, tumor-infiltrating T-cells, macrophages, and myeloid-derived suppressor cell (MDSCs)

Exploratory objective:

* To evaluate survival of patients treated with triplet combination regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age at time of screening
2. Patients must have histologic confirmation of MTAP-deficient metastatic urothelial carcinoma. MTAP-deficiency must be verified by institutional CLIA-certified IHC or by Next gen sequencing (such as FoundationOne or MDACC genomic analysis) showing copy number loss of MTAP gene. Histological variants such as glandular, squamous, sarcomatoid, micropapillary, plasmacytoid, and small cell changes will be allowed for this trial if these tumors are MTAP-deficient.
3. Patients can be considered for second line of therapy or beyond (after ICI with PD-(L)1 agent). Any prior intravesical therapy is allowed and does not count as a prior line of therapy.
4. All patients must have measurable disease by RECIST v1.1 and tumors of sufficient sizes for biopsy. In general, liver and lung lesions should be at least 1.0 cm, and patients with lymph node-only disease should have lesions of ≥ 1.5 cm in shortest dimension.

   Patients with disease confined to bone may be eligible if a measurable lytic defect is present. The study PI is the final arbiter in questions related to measurability. Patients with a three-dimensional mass or pelvic sidewall fixation on bladder examination under anesthesia are considered to have measurable disease.
5. Patients must have an ECOG performance status ≤ 2.
6. Adequate liver function as defined by AST or ALT ≤ 2.5 x ULN, or ≤ 5 x ULN if documented liver metastases are present.
7. Total bilirubin ≤ 1.5 x ULN, except subjects with Gilbert's syndrome or liver metastases, who must have a baseline total bilirubin ≤ 3.0 mg/dL.
8. Adequate bone marrow reserves as define by an ANC ≥ 1.5 x 109/L, hemoglobin ≥ 9 g/dL (may have been transfused), and platelets ≥ 100 x 109/L.
9. Adequate renal function as defined by a normal serum creatinine, or a creatinine clearance ≥ 45 ml/min [either measured using a 24 hour urine, calculated using CockroftGault, or estimated using the MDRD method from the National Kidney Disease Education Program (NKDEP) (the method reported by MDACC laboratories)] Cockroft-Gault formula: CrCl = [(140-age) • wt(kg)]/[72 •Creat (mg/dL)] (Multiply by 0.85 for females)
10. Negative serum or urine pregnancy test at screening for women of child-bearing potential.
11. Female participants of reproductive potential, defined as not surgically sterilized and between menarche and 1 year post menopause, must have a negative serum pregnancy test within 4 weeks prior to initiation of study treatment
12. Female participants of reproductive potential and male participants with female partners of reproductive potential must remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive measures from the start of study treatment until 30 days after the last dose of etrumadenant, 90 days after the last dose of zimberelimab, 180 days after the last dose of pemetrexed, whichever is longer.

    Please refer to appendix 5
13. The ability to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Pemetrexed. The ability to take folic acid, Vitamin B12, and dexamethasone according to protocol.

o. Mild autoimmune conditions (such as localized psoriasis or vitiligo) requiring minimal treatment or systemic autoimmune conditions well controlled by target agents such as an anti-IL-17 that do not affect overall immune system. Patients with a history of Hashimoto's thyroiditis only requiring hormone replacement, Type I diabetes, or conditions not expected to recur in the absence of an external trigger are allowed to participate.

p. Prior anti-PD-1/PD-L1 therapy is mandatory

Exclusion Criteria:

1. QTc ≥480 msec using Fredericia's QT correction formula
2. Due to the potential risk for drug-drug interactions with etrumadenant, participants must not have had:

a. Treatment with known BCRP substrates with a narrow therapeutic window, administered orally (e.g., prazosin, rosuvastatin) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of and throughout study treatment b. Treatment with known P-gp substrates with a narrow therapeutic window, administered orally (e.g., digoxin) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment c. Treatment with known strong CYP3A4 inducers (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort) and strong CYP3A4 inhibitors (e.g., clarithromycin, grapefruit juice, itraconazole, ketoconazole, posaconazole, telithromycin, and voriconazole) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment d. Refer to the following for more examples of relevant substrates, inhibitors, and inducers with the potential for drug-drug interactions with etrumadenant: https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-druginteractions-table-substrates-inhibitors-and-inducers

c. Any gastrointestinal condition that would preclude the use of oral medications (e.g., difficulty swallowing, nausea, vomiting, or malabsorption)

d. Prior treatment with an agent targeting the adenosine pathway

e. History of severe allergic reactions to chimeric or humanized antibodies or fusion proteins

f. Primary central nervous system (CNS) malignancies or CNS metastases, including leptomeningeal metastases, are not allowed. Subjects with previously treated brain metastases will be allowed if the brain metastases have been stable for at least 4 weeks following prior treatment and no ongoing steroid requirement.

g. Any other malignancy from which the patient has been disease-free for less than 2 years, except for non-melanomatous skin cancer, controlled localized prostate cancer, controlled thyroid papillary carcinoma, and in situ carcinoma of any site.

h. Women who are pregnant or breastfeeding or intend to become pregnant during their participation in the study.

i. Presence of large third space fluid which cannot be controlled by drainage. For patients who develop or have baseline clinically significant pleural or peritoneal effusions (on the basis of symptoms or clinical examination) before or during initiation of Pemetrexed therapy, consideration should be given to draining the effusion prior to dosing. However, if, in the investigator's opinion, the effusion represents progression of disease, the patient should be discontinued from study therapy.

j. Patients with active inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study.

k. Any condition requiring systemic treatment with corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids, steroids as premeds for hypersensitivity reactions, and adrenal replacement steroids doses ≤10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

l. History of primary immunodeficiency.

m. Patients who have prior organ transplantation, including allogeneic stem-cell transplant.

n. Live vaccinations within 4 weeks of the first dose of therapy and while on trials is prohibited. Receiving a COVID-19 vaccine at any timepoint will not result in exclusion from the trial.

o. True positive test results for active hepatitis A, B, or C during screening.

p. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

q. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, current pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrhythmia, or interstitial lung disease.

r. Uncontrolled psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.

s. Known allergy or hypersensitivity to study drug formulations.

t. Major surgical procedure (as defined by the PI or co-PIs within 28 days prior to the first dose of therapy) or still recovering from prior surgery.

u. Patient currently on dialysis.

v. Patients who had to discontinue checkpoint therapy due to grade 4 toxicity in the past

w. Prior antifolate therapy in the context of neoadjuvant chemotherapy or metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 and Number of Participants With Complete or Partial Response as their Best Overall Response per RECIST v1.1. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Omar Alhalabi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org